CLINICAL TRIAL: NCT00221494
Title: Can Additional Drug Therapy Accelerate Response Time to Antidepressants: A Double-blind, Placebo-controlled Randomization Research Study for Major Depression
Brief Title: Can Additional Drug Therapy Accelerate Response Time to Antidepressants
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI move
Sponsor: Mark Frye (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor-Investigator, Mark Frye, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 00-09-045-11
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2006-06

CONDITIONS: Depression
Keywords: depression
MeSH Terms: conditions — Depression | interventions — Citalopram; Pindolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: citalopram + tiodothyronine, or + pindolol, or + placebo

SUMMARY:
Antidepressants are commonly prescribed and are effective for treating depression. However, they generally take 4-6 weeks for a therapeutic response. This study is evaluating whether simultaneous treatment with thyroid hormone or pindolol can decrease the response time ("getting better faster") in patients who are starting SSRI treatment.

DETAILED DESCRIPTION:
Major depression is an illness with substantial personal and economic morbidity (Greenberg et al.1993) and antidepressants are the cornerstone of treatment. As antidepressants usually require 3-6 weeks of use before a response occurs, an effective antidepressant acceleration strategy would reduce the time of onset for an effective antidepressant response. This has significant clinical implications, as it could lead to reduced symptom morbidity, potentially reduce health care cost (i.e. shorter hospital length of stay), and improve functional capacity and quality of life.

The goal of this study is to enhance our understanding of strategies that accelerate or produce a more rapid treatment response in depression. This could lead to reduced symptom morbidity, potentially reduce health care cost (i.e. shorter hospital length of stay), and improve functional capacity and quality of life.

The study goals are: 1.) To assess whether the simultaneous commencement of liothyronine or pindolol to an SSRI can accelerate the treatment response (i.e. faster rate of improvement), 2.) To assess whether the simultaneous commencement of liothyronine or pindolol to an SSRI can augment or enhance treatment response (i.e. greater reduction in depressive symptoms at end of study phase), adn 3.) To assess whether gender influences the acceleration of augmentation response rate of liothyronine or pindolol.

ELIGIBILITY:
Inclusion Criteria:

1. Patients, male and female, between the ages of 18 to 65
2. DSM-IV criteria for major depressive disorder
3. No prior SSRI medication treatment (if a patient has discontinued a non-SSRI medication for side effects, they will not be excluded)
4. Ability to be followed clinically for 6 weeks
5. Each patient must understand the nature of the study and must sign an informed consent form

Exclusion Criteria:

1. Severe suicidality (as defined by Beck Depression Inventory Question 9, responses 2 or 3)
2. Major Axis I mental illness other than major depressive disorder
3. Unstable medical health specifically cardiovascular disease, abnormal EKG, history of severe drug allergy, poorly controlled diabetes, and asthma (pindolol contraindication)
4. History of thyroid disease or abnormal TFT's (stage I or II)
5. Need for adjunctive antipsychotic use or additional benzodiazepine during the study
6. Pregnancy
7. Seizure disorder
8. A positive urine toxicology screen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-01; Primary Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Frye, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Neuropsychiatric Institute, Los Angeles, California, United States